CLINICAL TRIAL: NCT06259175
Title: Evaluation of the Antihypertensive effectIveness, Tolerability, and Adherence With Amlodipine/ Indapamide/ Perindopril Triple Single-pill Combination in Hypertensive Patients Without Concomitant Antihypertensive Therapy (TRIPTYCH)
Acronym: TRIPTYCH
Status: Completed | Type: Observational
Sponsor: Servier Russia (Industry)
Responsible Party: Sponsor
Other Study IDs: IC4-06593-082-RUS
Record Dates: First submitted 2024-02-06; First posted 2024-02-14 (Actual); Last update posted 2025-06-11 (Actual); Status verified 2025-06

CONDITIONS: Arterial Hypertension; HTN
MeSH Terms: conditions — Hypertension | interventions — Amlodipine; Indapamide; Perindopril

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Amlodipine 5 mg + indapamide 1.25 mg + perindopril 5 mg — a triple fixed combination of Amlodipine , indapamide and perindopril combinations, was in a 3-month in accordance to the instruction for medical use approved in the Russian Federation
Drug: Amlodipine 5 mg + indapamide 2.5 mg + perindopril 10 mg — a triple fixed combination of Amlodipine , indapamide and perindopril combinations, was in a 3-month in accordance to the instruction for medical use approved in the Russian Federation
Drug: Amlodipine 10 mg + indapamide 2.5 mg + perindopril 10 mg — a triple fixed combination of Amlodipine , indapamide and perindopril combinations, was in a 3-month in accordance to the instruction for medical use approved in the Russian Federation

SUMMARY:
This is a multi-centre, observational, ambispective study, which will retrospectively and prospectively collect clinical and socio-demographic data from medical records of outpatients with arterial hypertension (HTN) initiated with the amlodipine/indapamide/perindopril SPC in real clinical settings.

375 patients to be included in the study in order for at least 300 patients to complete the study and provide an estimated 90% power of the study.

75 outpatient general practitioners and cardiologists will participate in this study.

DETAILED DESCRIPTION:
Patients will be managed in accordance with medical standards and clinical guidelines implemented in routine clinical practice. Once a patient is included in the study there will be 2 more additional visits scheduled for assessment of a patient's hemodynamic parameters as well as his/ her eligibility to continue to participate in the study, quality of life and treatment adherence statuses as well as presence or absence of adverse events. Second visit (V2) will be taking place approximately 8 weeks (± 1 week) after the date of the SPC initiation, visit V3 will be taking place approximately 12 weeks (± 1 week) after the date of the SPC initiation.

ELIGIBILITY:
Inclusion Criteria:

* Obtained signed informed consent from the patient.
* Patients of 18 years and older.
* Treatment with the amlodipine/indapamide/perindopril SPC in accordance with the Summary of Product Characteristics (SmPC) approved for medical use in the Russian Federation (RF) (Arterial hypertension - SBP ≥ 140 mm Hg and/or DBP ≥ 90 mm Hg), for a period of 2 to 4 weeks at the time of inclusion in the study.
* Absence of any other additional antihypertensive medical treatment with β-blockers, α-blockers, I1-imidazoline receptor agonists, loop and potassium-sparing diuretics from the initiation of the SPC to the inclusion visit (V1).
* Clinical parameters of the primary interest (resting SBP and DBP) are available in medical records for the nearest date before the initiation of the amlodipine/indapamide/perindopril SPC.

Exclusion Criteria:

* Subjects who are unwilling or unable to provide a signed Informed Consent Form.
* Any contraindication to the treatment with the amlodipine/indapamide/perindopril SPC according to its' approved SmPC for medical use in RF.
* Presence of indications for concomitant therapy with β-blockers, α-blockers, I1-imidazoline receptor agonists, loop and potassium-sparing diuretics.
* Expected poor adherence to the administration of the prescribed SPC due to patient's lack of co-operation that according to the physician's opinion, is likely to jeopardize the interaction between the patient and the investigator during the study.
* Any severe, decompensated or unstable somatic diseases or conditions that according to investigator discretion are life-threatening or worsen the prognosis for the patient: stroke/TIA, myocardial infarction or unstable angina occurred within 3 months before the inclusion date, angina pectoris IV functional class, chronic heart failure IV functional class by NYHA, current decompensation of diabetes mellitus, autoimmune or oncological diseases, severe or chronic poorly controlled cardiac arrhythmias, gastrointestinal disorders affecting absorption, severe hepatic diseases, pancreatic diseases, severe allergic reactions, connective tissue diseases etc.
* Secondary arterial hypertension.
* Alcohol or any drug abuse.
* Surgical interventions on heart or coronary vessels (i.e., heart valve replacement, stent implantation or CABG), or any non-cardiological serious surgical intervention that are planned within next 3 months and may require withdrawal or changes in current therapy.
* Participating in any other clinical trial currently or for 30 days period before informed consent was signed.
* Patient's decision to withdraw from the study due to any reasons.
* Any contraindication to the treatment with the amlodipine/indapamide/perindopril SPC according to its' approved SmPC for medical use in RF occurred during the follow-up period.
* Clinical situation(s) requiring adding to the SPC other CV medicines such as β-blockers, α-blockers, I1-imidazoline receptor agonists, diuretics, calcium antagonists and/or ACE inhibitors.
* Clinical situation(s) requiring withdrawing the SPC from the treatment scheme of a patient.
* Uncooperative patient's behavior resulting, upon investigating physician's opinion, in resolute unwillingness of the patient to collaborate with the physician therefore jeopardizing effectiveness of the entire treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: outpatients with arterial hypertension (HTN) who do not receive any other concomitant antihypertensive medicines within 12 weeks from the initiation of the SPC.
Sampling Method: Non-Probability Sample
Enrollment: 396 (Actual)
Dates: Start 2024-05-01 (Actual); Primary Completion 2025-04-21 (Actual); Study Completion 2025-06-01 (Actual)

PRIMARY OUTCOMES:
To describe antihypertensive effectiveness of the triple single-pill combination (SPC) of amlodipine, indapamide and perindopril in outpatients with arterial hypertension (HTN) who do not receive any other concomitant antihypertensive medicines within 12 | 12 weeks
  Mean changes from baseline (BL) in SBP (systolic blood pressure) assessed at V3 (12+1 weeks after the SPC initiation).
To describe antihypertensive effectiveness of the triple single-pill combination (SPC) of amlodipine, indapamide and perindopril in outpatients with arterial hypertension (HTN) who do not receive any other concomitant antihypertensive medicines within 12 | 12 weeks
  Mean changes from baseline (BL) in DBP (diastolic blood pressure) assessed at V3 (12+1 weeks after the SPC initiation).

SECONDARY OUTCOMES:
To describe changes in systolic blood pressure (SBP) from baseline to weeks 4 and 8 from the SPC initiation. | 4 weeks
  Mean change from BL in SBP assessed at V1 (4+1 weeks after the SPC initiation)
To describe changes in diastolic blood pressure (DBP) from baseline to weeks 4 and 8 from the SPC initiation. | 4 weeks
  Mean change from BL in DBP assessed at V1 (4+1 weeks after the SPC initiation)
To describe changes in systolic blood pressure (SBP) from baseline to weeks 4 and 8 from the SPC initiation. | 8 weeks
  Mean change from BL in SBP assessed at V2 (8+1 weeks after the SPC initiation).
To describe changes in diastolic blood pressure (DBP) from baseline to weeks 4 and 8 from the SPC initiation. | 8 weeks
  Mean change from BL in SBP and DBP assessed at V2 (8+1 weeks after the SPC initiation).
To describe a proportion of patients who reached SBP target goals at week 12 from the SPC initiation. | 12 weeks
  Proportion of patients who reached SBP ≤130 mm Hg at V3 (12+1 weeks after the SPC initiation).
To describe a proportion of patients who reached DBP target goals at week 12 from the SPC initiation. | 12 weeks
  Prortion of patients who reached DBP <80 mm Hg at V3 (12+1 weeks after the SPC initiation).
To describe changes in patients' quality-of-life throughout the observational period of the study. | 12 weeks
  Mean changes in scores of the Health-related quality of life Questionnaire for Patients with Hypertension (HRQoL) assessed at V3 (12+1 weeks after the SPC initiation).

CONTACTS AND LOCATIONS:
Overall Officials: Alexandra Konradi, Principal Investigator — Medical Education Institute
Locations (1):
- Servier, Moscow, Russia